CLINICAL TRIAL: NCT02714530
Title: Concomitant Radiotherapy and Erlotinib in Advanced Lung Cancer
Brief Title: Thoracal Radiotherapy and Tarceva
Acronym: ThoRaT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Åslaug Helland, MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ThoRaT
Record Dates: First submitted 2015-09-10; First posted 2016-03-21 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Erlotinib Hydrochloride; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy combined with erlotinib (Experimental): Standard treatment 3 Gy x 10 to lung tumor and mediastinal lymph nodes and erlotinib given concomitantly, 150 mg p.o. daily from the day before radiation, until the last day of radiation.
  Interventions: Drug: Erlotinib; Radiation: Radiation
- Radiotherapy alone (Active Comparator): Radiotherapy 3 Gy x 10 alone
  Interventions: Radiation: Radiation

INTERVENTIONS:
Drug: Erlotinib — Tarceva daily during radiotherapy course
  Other Names: Tarceva
  Arms: Radiotherapy combined with erlotinib
Radiation: Radiation — Radiotherapy

SUMMARY:
The purpose of this study is to determine if erlotinib given orally along with concurrent palliative irradiation to lung cancer improves local control compared to those treated with radiotherapy alone.

DETAILED DESCRIPTION:
Endpoints:

Primary:

* To determine if erlotinib given orally along with concurrent external beam radiation therapy, prolongs local tumour control as determined by CT evaluation compared to treatment with external beam radiation therapy alone

Secondary:

* To confirm the safety profile of erlotinib along with concurrent external beam radiation therapy.
* To evaluate if erlotinib along with concurrent external beam radiation therapy, improve quality of life as assessed with the EORTC QLQ-C30 and the EORTC QLQ-LC13.
* To evaluate if PET-CT examination can be used to predict response to treatment.
* To evaluate overall survival in the different groups

Trial Design: Open multicenter two-armed randomized phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Histological or cytological verified NSCLC
* Palliative radiotherapy to thorax indicated
* ECOG Performance status 0-2
* Fertile patients must use contraception
* Signed informed consent
* Ability to understand and fill in QoL questionnaires
* Capability to take per os medication
* Serum bilirubin < 2 times upper limit of normal (ULN)
* AST and ALT < 2 times ULN (< 5 times ULN if liver metastases are present)
* Creatinine < 5 times ULN

Exclusion Criteria:

* Pregnancy or nursing
* Other prior or concurrent malignant disease likely to interfere with study treatment or comparisons
* No evidence of other significant laboratory finding or concurrent uncontrolled medical illness, that in the opinion of the investigator, would interfere with study treatment or results comparison or render the patient at high risk for treatment complications
* No prior radiotherapy to the same organ / place
* No concurrent treatment with other experimental drugs
* Known brain metastases in need of radiotherapy
* Known hypersensitivity to erlotinib or other substances in the erlotinib tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with progression in radiation field among patients treated with erlotinib combined with radiotherapy compared to radiotherapy alone | 1 year
  Evaluate local control by radiological evaluation

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events grade >3 as Assessed by CTCAE v4.0 | 1 year
  To confirm the safety profile of erlotinib along with concurrent external beam radiation therapy.
Overall survival will be measured | 1 year
  To evaluate overall survival in the different groups

CONTACTS AND LOCATIONS:
Overall Officials: Åslaug Helland, MD PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo, International/Other
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
Publish results

REFERENCES:
- [Derived] Nymoen HM, Alver TN, Horndalsveen H, Eide HA, Bjaanaes MM, Brustugun OT, Gronberg BH, Haakensen VD, Helland A. Thoracic radiation in combination with erlotinib-results from a phase 2 randomized trial. Front Oncol. 2024 Aug 1;14:1412716. doi: 10.3389/fonc.2024.1412716. eCollection 2024. PMID 39148905
- [Derived] Abravan A, Eide HA, Londalen AM, Helland A, Malinen E. Mapping Bone Marrow Response in the Vertebral Column by Positron Emission Tomography Following Radiotherapy and Erlotinib Therapy of Lung Cancer. Mol Imaging Biol. 2019 Apr;21(2):391-398. doi: 10.1007/s11307-018-1226-7. PMID 29916117